CLINICAL TRIAL: NCT04884594
Title: Intravenous Administration of AAV8-human Cocaine Hydrolase to Treat Cocaine Use Disorder
Brief Title: AAV8-hCocH for Cocaine Use Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: W. Michael Hooten (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, W. Michael Hooten, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 20-012225; 5UH3DA042492 (NIH)
Record Dates: First submitted 2021-05-07; First posted 2021-05-13 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Cocaine Dependence, in Remission
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- AAV8-hCocH dose level 1: 2e12 vg/kg (Experimental): Cohort 1: Participant receives one-time IV administration of low dose 2e12 vg/kg of AAV8-hCocH, with 7 week of follow-up after dose
  Interventions: Drug: AAV8-hCocH
- AAV8-hCocH dose level 3: 6e12vg/kg (Experimental): Cohort 3: Participant receives one-time IV administration of medium dose 6e12vg/kg of AAV8-hCocH, with 7 week of follow-up after dose
  Interventions: Drug: AAV8-hCocH
- AAV8-hCocH dose level 2: 4e12vg/kg (Experimental): Cohort 2: Participant receives one-time IV administration of medium dose 4e12vg/kg of AAV8-hCocH, with 7 week of follow-up after dose
  Interventions: Drug: AAV8-hCocH

INTERVENTIONS:
Drug: AAV8-hCocH — 2e12 vg/kg single infusion intravenous
  Arms: AAV8-hCocH dose level 1: 2e12 vg/kg
Drug: AAV8-hCocH — 6e12 vg/kg single infusion intravenous
  Arms: AAV8-hCocH dose level 3: 6e12vg/kg
Drug: AAV8-hCocH — 4e12 vg/kg single infusion intravenous
  Arms: AAV8-hCocH dose level 2: 4e12vg/kg

SUMMARY:
The purpose of this study is to test the safety of a novel gene viral vector treatment for adults with cocaine use disorder-sustained remission. This gene regulates an enzyme (cocaine hydrolase) that breaks down cocaine into inactive substances, thereby decreasing the pleasurable feeling this drug usually provides.

DETAILED DESCRIPTION:
This is a phase-I dose escalation clinical trial testing the safety and MTD of IV administration of AAV8-hCocH to subjects with a history of cocaine use disorder-sustained remission. Subjects who provide written informed consent, meet entry criteria, and do not have transduction inhibition to AAV8 (pre-existing AAV8 antibodies) will be eligible. Subjects will be enrolled sequentially every 2-3 months or longer between cohorts. Dose escalation may be initiated after a single subject has been safely dosed; maximum enzyme expression is anticipated at week 3-4. This escalation paradigm is intended to minimize the number of subjects exposed to sub-therapeutic doses. The starting dose is based on the expression and safety of AAV8-CocH in mice, rats and NHP, and previous human experience using AAV8-FVIII IV in hemophilia patients. The starting dose has a large safety margin (15-fold) from the NOAEL in NHP. Approximately 7 weeks after an injection, a decision to escalate to the next dose level will be made based on a review of safety parameters and CocH levels by the investigative team.

ELIGIBILITY:
Inclusion Criteria:

* Non-treatment seeking male or females ages 18 to 65 years, inclusive.
* DSM-5 diagnosis of cocaine use disorder in sustained remission as confirmed by the PI's review of the medical record.
* Are motivated to abstain from cocaine use during the period of the study, as evidenced both by the judgment of the Investigator or designee and by compliance with the requirement to make regular clinic visits.
* In the opinion of the PI, be in good general health as determined by medical and psychiatric history, general clinical examination, vital signs, and laboratory tests.
* Have provided written informed consent. Subjects should be cooperative, willing and able to participate and adhere to the protocol requirements.
* Have hematology, chemistry, kidney and liver function laboratory tests that are within (+/- 10%) of the current Mayo Clinic standardized normal values.
* Show a baseline EKG that demonstrates normal sinus rhythm and conduction without clinically significant abnormalities or arrhythmias.
* Are willing to return to research area for follow-up.

Exclusion Criteria:

* They show detectable pre-existing immunity to the AAV8 capsid as measured by AAV8 transduction inhibition and AAV8 total antibodies.
* Evidence of HIV or hepatitis of any etiology.
* Creatinine ≥ 1.5 mg/dL.
* Any disease or mental health condition at the physician's discretion that would prevent the subject from fully complying with the requirements of the study. The physician may exclude subjects with active alcohol abuse, other substance abuse or positive urine toxicology screen for substances of abuse.
* Pregnant &/or lactating. All lactating women will be excluded from study participation. Women of child-bearing potential must have a negative pregnancy test performed at screening visit, agree to use birth control throughout the study period, refrain from getting pregnant within the study period and consent to pregnancy testing throughout the study period. Men must agree to use barrier methods of birth control and refrain from fathering children within the next year.
* Morbid obesity (BMI > 40).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 60 months
  Number of participants with treatment-related adverse events
Change in enzyme expression profile | Baseline, 24 months
  Serum level of AAV8-hCocH gene expression

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 24 months
  Cmax is measured as the peak concentration of AAV8 in the blood after intravenous infusion
Time of peak concentration (tmax) | 24 months
  The time to maximum plasma concentration of AAV8 in the blood after intravenous infusion
Half-Life (t1/2) | 24 months
  The time for plasma concentration of AAV8 in the blood to be reduced to exactly half of starting concentration
Area under the Concentration-Time Curve (AUC) | 24 months
  AUC is a measure of the AAV8 serum concentration over time. Used to characterize drug absorption.

CONTACTS AND LOCATIONS:
Overall Officials: W. Michael Hooten, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No